CLINICAL TRIAL: NCT01731860
Title: Pilot Study Intended to Provide Input for Future Designs Using the PET Alpha Ring Detector and to Support the Pre-market Notification of a Future Product
Brief Title: Pilot Study Intended to Provide Input for Future Designs Using the PET Alpha Ring Detector
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Collaborators: University Hospitals Cleveland Medical Center (Other); Case Western Reserve University (Other); Imarc Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Alpha Ring 12-001
Record Dates: First submitted 2012-11-09; First posted 2012-11-22 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Focus of Study is Imaging Performance With the New Technology Compared With the Currently Available Technology.
Keywords: PET/CT; Philips

ARMS (1):
- Patients receiving PET/CT (Experimental): Patients already scheduled for a clinically necessary PET/CT scan.
  Interventions: Device: Additional PET Scan

INTERVENTIONS:
Device: Additional PET Scan — Additional PET Scan with no additional radiopharmaceutical administration.

SUMMARY:
A standard PET/CT scanner is comprised of two different machines: An X-ray computed tomography scanner (CT), which gives information about your anatomy, and a Positron Emission Tomography scanner (PET) that provides information about how the body functions. Both of these work together to make the final images for doctors to review. As part of this research study the investigators would like to test a new scanner technology by evaluating the quality of the images obtained using this new PET system.

The scanner the investigators would use is able to do both types of examination, the standard PET/CT and the additional research PET. The new PET system adds a second scanner ring to the standard PET/CT. This allows the patient to stay on the same imaging table for both studies. Being in this study does not change how the standard PET/CT will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients are at least 18 years
* Patients are medically stable
* Patients scheduled for clinically necessary PET/CT examination

Exclusion Criteria:

* Patients who are pregnant
* Patients who are unwilling/unable to sign the Informed Consent Form
* Patients who are cognitively impaired and unable to provide informed consent
* Patients who have experienced adverse events to PET/CT examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-11; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Imaging Capabilities and Performance of the Alpha Ring | Within 1 month of image acquisition
  Images acquired using the investigational device will be compared with the images obtained using the approved clinical device. The qualitative image review will be performed by the reading radiologist/nuclear medicine physician.

CONTACTS AND LOCATIONS:
Overall Officials: Peter F Faulhaber, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospital Case Medical Center, Cleveland, Ohio, United States